CLINICAL TRIAL: NCT03854786
Title: A Randomized, Placebo-controlled, Multi-blind Study to Assess the Effect of Oxyjun on Aerobic Fitness in Overweight and Obese Individuals.
Brief Title: Aerobic Fitness in Overweight and Obese Individuals
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to Covid - 19 pandemic
Sponsor: Vedic Lifesciences Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: EB/181201/OXYJUN/EVRG
Record Dates: First submitted 2019-02-21; First posted 2019-02-26 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2020-01

CONDITIONS: Healthy
MeSH Terms: interventions — PACEBO protocol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oxyjun (Active Comparator): Oxyjun- 400 mg OD after breakfast
  Interventions: Dietary Supplement: Oxyjun
- Methyl Crystalline Cellulose (Placebo Comparator): Methyl Crystalline Cellulose- 400 mg OD after breakfast
  Interventions: Dietary Supplement: Pacebo

INTERVENTIONS:
Dietary Supplement: Oxyjun — Oxyjun is the proprietary single ingredient product containing high concentrated well standardized aqueous extract of Terminalia arjuna.
  Arms: Oxyjun
Dietary Supplement: Pacebo — Methyl Crystalline Cellulose
  Arms: Methyl Crystalline Cellulose

SUMMARY:
Oxyjun is known for improving cardiovascular endurance. Overweight and obese individuals are at increased risk of cardiovascular complications. To lower the risk, these individuals need to remain physically active with acceptable aerobic fitness.

Hence, the objective of the study is to investigate the effect of Oxyjun on aerobic fitness in physically active overweight and obese individuals. All subjects in the study will be tested for maximum aerobic capacity , body composition, and serum biomarker for fitness.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index ≥ 25 - ≤ 34.9 kg/m2.
* Waist Circumference ≥ 80 cms.
* Non-smoker.
* BP ≤ 140/90 mm Hg
* FBS ≤ 125 mg/dl
* Hb ≥ 11 g/ dl
* Can abstain from strenuous exercise and alcohol for at least 48 hours.
* Can abstain from caffeine for at least 24 hours.

Exclusion Criteria:

* Participants with history of regular (≥2 times a week) structured exercise (gym, walking, yoga, etc).
* Inter-arm blood pressure is ≥10 mm Hg.
* Known cases of type II Diabetes Mellitus.
* Known cases of hypertension with or without anti-hypertensive medication.
* Visual or balance problems, or who cannot walk on a treadmill without using the handrails.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 11 (Actual)
Dates: Start 2020-01-03 (Actual); Primary Completion 2020-03-05 (Actual); Study Completion 2020-05-28 (Actual)

PRIMARY OUTCOMES:
To investigate the effect on Oxyjun on aerobic fitness in overweight and obese individuals | From baseline to Day 56
  Measured by change in VO2 max

CONTACTS AND LOCATIONS:
Locations (1):
- Vedic Lifesciences Pvt. Ltd, Mumbai, Opp Infinity Mall, India